CLINICAL TRIAL: NCT06021717
Title: PCA Ketamine-Morphine Versus PCA Morphine as Post-Operative Analgesia in Colorectal Surgery
Brief Title: PCA Ketamine-Morphine VS PCA Morphine as Post-Operative Analgesia in Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JEP-2018-092
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-05

CONDITIONS: Ketamine; Morphine
Keywords: Colorectal surgery; patient-controlled analgesia; postoperative pain management
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated into either Group A or Group B by computer-generated randomization a day before planned surgery.
  Group A will receive PCA ketamine-morphine 0.5 mg/ml in 1:1 ratio while group B will receive PCA morphine 1mg/ml,
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients, nurses who cared for the patients, the anesthetist who performed the anesthesia and the investigators who gathered the data were blinded to patients' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): PCA ketamine (Ketamine HCl, Pfizer Inc., US) 0.5 mg plus morphine 0.5 mg ml-1 (ratio 1:1) as postoperative analgesia.
  Interventions: Drug: Ketamine-Morphine
- Group B (Active Comparator): PCA morphine (Pfizer Inc., US) 1 mg ml-1 as postoperative analgesia.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine-Morphine — PCA ketamine (Ketamine HCl, Pfizer Inc., US) 0.5 mg plus morphine 0.5 mg ml-1 (ratio 1:1)
  Other Names: Ketamine Hydrochloric, Pfizer Inc., US; Morphine Pfizer Inc., US
  Arms: Group A
Drug: Morphine — PCA morphine (Pfizer Inc., US) 1 mg ml-1
  Other Names: Morphine Pfizer Inc., US
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of PCA ketamine-morphine versus conventional PCA morphine in postoperative patients undergoing elective laparotomy colorectal surgery under general anaesthesia. The specific objectives are:

1. To compare the post-operative analgesic requirement with PCA ketamine-morphine in comparison with PCA morphine.
2. To compare the postoperative pain scores between PCA ketamine-morphine and PCA morphine.
3. To assess patients' overall satisfaction with PCA ketamine-morphine in comparison with PCA morphine.
4. To study the incidence of side effects of PCA ketamine-morphine in comparison with PCA morphine.

Participants will be screened and recruited at pre-anaesthetic clinic (PAC). Those who consented will be taught to use PCA machine and the potential side effects of the study drugs. They will be randomly allocated into either Group A or Group B by computer generated randomization a day before planned surgery.

Researchers will compare Group A and Group B to see post-operative pain scores, patients' overall satisfaction and any incidence of side effects.

DETAILED DESCRIPTION:
INTRODUCTION

Patient-controlled analgesia (PCA) is an established, efficient and safe technique for providing postoperative analgesia and has been associated with better pain relief and patient satisfaction with less postoperative complications and side effects [1]. Despite years of advances in pain management, opioids have been the mainstay for treatment of postoperative pain particularly in moderate to severe pain. Of all opioids, morphine is the most studied drug and remains the drug of choice for PCA, especially in Malaysian hospitals. However, morphine usage is also associated with known side effects such as sedation, nausea and vomiting, pruritus, urinary retention and respiratory depression [2]. A review of 32 studies involving opioids-based PCA-22 of which were PCA morphine-reported an incidence of 19% nausea, 18.1% vomiting, 30.9 % of nausea and/or vomiting, 25.7% sedation, 17.9% urinary retention, 17.9% pruritus and 15.2% hypoxia and 1.6% respiratory depression that may be life-threatening associated with PCA opioids use [3, 4]. The concept of multimodal analgesia hence was introduced to reduce opioid-related side effects. Adjuvants such as acetaminophen and non-steroidal anti-inflammatory drugs are commonly used nowadays in combination with opioids as opioid-sparing agents to reduce opioid usage [5].

Ketamine, an N-methyl-D-aspartate (NMDA) antagonist, has undergone a recent resurgence of interest among acute care providers as an adjunct in acute pain management [6, 7]. Ketamine at a sub-anesthetic dose (0.2-0.5 mg kg-1) produces intense analgesia [5, 8]. Since its development in 1962, various studies have been conducted to prove the efficacy of ketamine as post-operative analgesia and as an opioid-sparing agent [8-10]. A review by Laskowski and colleagues described that IV ketamine improved the quality of pain control, in addition to decreased opioid consumption with the particular benefit being observed in painful procedures, such as upper abdominal, thoracic, and major orthopedic surgeries [11]. While Carstensen and co-workers in a qualitative review comparing PCA ketamine-morphine with PCA morphine alone also described the superior efficacy of ketamine-morphine in providing pain control with a significantly higher incidence of opioid-related side effects in the morphine group [12]. In comparison to opioids, ketamine's lack of respiratory depressant effects also favors its use as an opioid adjunct in patients with airway and respiratory compromise, especially in morbid obesity and post-thoracotomy patients [13, 14].

Despite the potential efficacy with published evidence of PCA ketamine-morphine in postoperative pain management, its use is not well established in most Malaysian hospitals including the current study site. Hence, the aim of this study was to evaluate the effectiveness of PCA ketamine-morphine in comparison to conventional PCA morphine alone as postoperative analgesia in colorectal surgery patients in the current study site.

METHODS

This prospective double-blind randomized controlled trial was conducted in Hospital Sultanah Aminah Johor Bahru from February to October 2018 after obtaining ethics approval from the local and institutional ethics committee (NMRR-17-1863-37291 & JEP-2018-092). Sixty elective American Society of Anaesthesiologists (ASA) I or II patients scheduled for lower midline laparotomy colorectal surgery aged between 18-70 years old were recruited and informed consents were obtained. Patients with a known allergy to morphine or ketamine, uncontrolled hypertension, past history of chronic pain on regular analgesics, psychiatric illness on psychiatric drugs, BMI more than 35 and creatine clearance less than 30 were excluded from the study. All patients who consented were taught the usage of a PCA machine and the potential side effects of ketamine and morphine preoperatively. They were randomly allocated into either Group A or Group B by computer-generated randomization a day before planned surgery.

Group A received PCA ketamine (Ketamine HCl, Pfizer Inc., US) 0.5 mg plus morphine 0.5 mg ml-1 (ratio 1:1) while Group B received PCA morphine (Pfizer Inc., US) 1 mg ml-1 as postoperative analgesia. There was no baseline infusion and the lock-out period was set to 5 minutes. The study drugs were prepared one day before the surgery by the pharmacist who was not involved in the intraoperative and post-=operative management of the patients. The drugs were labelled as study drugs with the study number. The patients, nurses who cared for the patients, the anesthetist who performed the anesthesia and the investigators who gathered the data were blinded to patients' group allocation.

All patients had standard monitoring of blood pressure, electrocardiogram (ECG), oxygen saturation and end-tidal carbon dioxide (CO2). They were pre-oxygenated with 100% oxygen for 2-3 minutes. The induction of general anesthesia was standardized to intravenous (IV) fentanyl (Cephalon Inc., US) 2 mcg kg-1, IV propofol (Diprivan, Pfizer Inc., US) 2 mg kg-1 and IV rocuronium (US) 0.6 mg kg-1 and intubation with the appropriate size of the endotracheal tube. Anesthesia was maintained with desflurane (Suprane, Novartis AG, Switzerland) in a mixture of 50% of oxygen and 50% of air, and titrated to achieve a minimum alveolar concentration (MAC) of 1.0. All patients received IV dexamethasone (US) 8 mg after induction and IV morphine 0.1 mg kg-1 as intraoperative analgesia. Boluses of IV fentanyl 25 mcg were given if extra analgesia was required and recorded. IV ondansetron (US) 4 mg was given upon initiation of skin closure. The skin incision site was infiltrated with 0.25% Bupivacaine (US) 10-20 ml during skin closure. The standard dose of IV neostigmine and IV atropine was used to reverse residual neuromuscular blockade at the end of surgery.

At the recovery bay, pain score was assessed using the Numerical Rating Scale (NRS), by which patients scored their pain intensity between number 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable. If the pain score was > 4 at rest, IV morphine boluses were given and titrated according to the pre-set morphine protocol until the pain score was ≤ 4. PCA machine with the study drug(s) was commenced once the pain score was ≤ 4 at rest.

Patients were assessed 30 minutes after the commencement of PCA, at 6 hourly intervals for the first 24 hours and subsequently at 12 hourly intervals for the next 24 hours post-operatively by the Acute Pain Service (APS) team. They were solely on PCA as post-operative analgesia as the patients were kept nil by mouth for the first 48 hours postoperatively. All patients were assessed for pain score, sedation score, respiratory rate and other side effects of morphine and ketamine including nausea and vomiting, pruritus, dizziness and hallucinations. If the pain score was > 4 at rest during the assessment, 2 ml of PCA drug was given as boluses and titrated every 10 minutes to achieve a pain score ≤ 4.

Cumulative morphine consumption was also recorded. Sedation was assessed using Pasero Opioid-Induced Sedation Scale (POSS) (S - sleep, easy to arouse, 1 - awake and alert, 2 - slightly drowsy, easy to arouse, 3 - frequently drowsy, arousable, drift to sleep during the conversation, 4 - somnolent, minimal or no response to verbal or physical stimulation). Treatment for nausea, vomiting and pruritus was given as deemed appropriate and recorded. At 48-hour post-operation, the patient's overall satisfaction score was assessed using 1 to 5 Likert scale (1 - very unsatisfied, 2 - unsatisfied, 3 - neutral, 4 - satisfied and 5 - very satisfied). If patients experience hallucinations or delirium, PCA bolus dose was reduced by 0.2 ml and the symptoms were reassessed after 1 hour. If symptoms persist, the PCA bolus dose was reduced further by 0.2 ml every hour until symptoms disappear and PCA subsequently continued at the reduced dose.

Patients with complicated surgeries in which they became haemodynamically unstable and required post-operative ICU admission, developed anaphylaxis after commencement of study drugs, developed persistent delirium or hallucination after reduction of PCA bolus dose and pain was uncontrollable with the reduced dose or those who refused to continue with the study for any reasons were withdrawn from the study and given other means of analgesia as appropriate by the acute pain service (APS) team.

The sample size was calculated using 'Power and Sample Size Calculations' program. The sample size was estimated using t-test calculation as derived from mean pain score and standard deviation as quoted in a study by Javery and colleagues [15]. The α value was set at 0.05 and power of study at 90% and standard deviation at 1.67, whereby it was estimated that 27 patients were required for each group. Anticipating a 10% drop-out rate, 30 patients were eventually recruited in each group, resulting in 60 patients for the whole study.

All data were analyzed using the SPSS (Statistical Package for The Social Sciences) software. Chi-square test or Fisher exact test was used when appropriate to calculate any significant differences for categorical variables. Independent t-test or Mann Whitney U test was used as appropriate to determine any significant differences for continuous variables. The incidence of side effects between the two groups was compared using Chi-square test. A P value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Elective American Society of Anaesthesiologists (ASA) I or II patients scheduled for lower midline laparotomy colorectal surgery aged between 18-70 years old

Exclusion Criteria:

* Patients with a known allergy to morphine or ketamine, uncontrolled hypertension, past history of chronic pain on regular analgesics, psychiatric illness on psychiatric drugs, BMI more than 35 and creatine clearance less than 30.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
PCA drugs demanded and delivered | 30 minutes after commencement of PCA until 48 hours
  Total PCA drugs demanded and delivered
Pain score | 30 minutes after commencement of PCA until 48 hours
  Pain score at rest and on movement with NRS
  Numerical Rating Scale (NRS) for pain score assessment A numerical pain assessment tool from 0 to 10, where 0 denotes no pain, 5 denotes moderate pain and 10 denotes worst possible pain.
Incidence of side effects | 30 minutes after commencement of PCA until 48 hours
  * Opiod related side effects : nausea and vomiting, pruritus, dizziness, respiratory depression and treatment on PRN basis if indicated
  * Ketamine related side effects : delirium, hallucinations, hypertension, tachycardia
Patients' overall satisfaction | At 48 hours post oeprative
  Assessment of patients' overall satisfaction with a 5-points scales at 48 hours.
  A 5-point scale from 1 to 5, where:
  1. = very unsatisfied
  2. = unsatisfied
  3. = neutral
  4. = satisfied
  5. = very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Chian Yong Liu, MMed (Anaes), Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pouldar TM, Maher DP, Betz AW, Wiegers JJ, Friedman JA, Zaidi SS, Rejali A, Tran HP, Yumul R, Louy C. Adverse Effects Associated with Patient-Controlled Analgesia with Ketamine Combined with Opioids and Ketamine Infusion with PCA Bolus in Postoperative Spine Patients: A Retrospective Review. J Pain Res. 2022 Oct 10;15:3127-3135. doi: 10.2147/JPR.S358770. eCollection 2022. PMID 36247824
- [Background] Ragazzoni L, Kwizera A, Caviglia M, Bodas M, Franc JM, Ssemmanda H, Ripoll-Gallardo A, Della-Corte F, Alenyo-Ngabirano A. Intra-operative low-dose ketamine does not reduce the cost of post-operative pain management after surgery: a randomized controlled trial in a low-income country. Afr Health Sci. 2019 Dec;19(4):3127-3135. doi: 10.4314/ahs.v19i4.35. PMID 32127889
- [Background] Viderman D, Tapinova K, Nabidollayeva F, Tankacheev R, Abdildin YG. Intravenous versus Epidural Routes of Patient-Controlled Analgesia in Abdominal Surgery: Systematic Review with Meta-Analysis. J Clin Med. 2022 May 5;11(9):2579. doi: 10.3390/jcm11092579. PMID 35566705
- [Background] Walder B, Schafer M, Henzi I, Tramer MR. Efficacy and safety of patient-controlled opioid analgesia for acute postoperative pain. A quantitative systematic review. Acta Anaesthesiol Scand. 2001 Aug;45(7):795-804. doi: 10.1034/j.1399-6576.2001.045007795.x. PMID 11472277
- [Background] Argoff CE. Recent management advances in acute postoperative pain. Pain Pract. 2014 Jun;14(5):477-87. doi: 10.1111/papr.12108. Epub 2013 Aug 15. PMID 23945010
- [Background] Hansen KB, Yi F, Perszyk RE, Furukawa H, Wollmuth LP, Gibb AJ, Traynelis SF. Structure, function, and allosteric modulation of NMDA receptors. J Gen Physiol. 2018 Aug 6;150(8):1081-1105. doi: 10.1085/jgp.201812032. Epub 2018 Jul 23. PMID 30037851
- [Background] Simonini A, Brogi E, Cascella M, Vittori A. Advantages of ketamine in pediatric anesthesia. Open Med (Wars). 2022 Jul 6;17(1):1134-1147. doi: 10.1515/med-2022-0509. eCollection 2022. PMID 35859796
- [Background] Brinck ECV, Virtanen T, Makela S, Soini V, Hynninen VV, Mulo J, Savolainen U, Rantakokko J, Maisniemi K, Liukas A, Olkkola KT, Kontinen V, Tarkkila P, Peltoniemi M, Saari TI. S-ketamine in patient-controlled analgesia reduces opioid consumption in a dose-dependent manner after major lumbar fusion surgery: A randomized, double-blind, placebo-controlled clinical trial. PLoS One. 2021 Jun 7;16(6):e0252626. doi: 10.1371/journal.pone.0252626. eCollection 2021. PMID 34097713
- [Background] Zhou L, Yang H, Hai Y, Cheng Y. Perioperative Low-Dose Ketamine for Postoperative Pain Management in Spine Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Pain Res Manag. 2022 Mar 31;2022:1507097. doi: 10.1155/2022/1507097. eCollection 2022. PMID 35401887
- [Background] Wang L, Johnston B, Kaushal A, Cheng D, Zhu F, Martin J. Ketamine added to morphine or hydromorphone patient-controlled analgesia for acute postoperative pain in adults: a systematic review and meta-analysis of randomized trials. Can J Anaesth. 2016 Mar;63(3):311-25. doi: 10.1007/s12630-015-0551-4. Epub 2015 Dec 10. PMID 26659198
- [Background] Laskowski K, Stirling A, McKay WP, Lim HJ. A systematic review of intravenous ketamine for postoperative analgesia. Can J Anaesth. 2011 Oct;58(10):911-23. doi: 10.1007/s12630-011-9560-0. Epub 2011 Jul 20. PMID 21773855
- [Background] Carstensen M, Moller AM. Adding ketamine to morphine for intravenous patient-controlled analgesia for acute postoperative pain: a qualitative review of randomized trials. Br J Anaesth. 2010 Apr;104(4):401-6. doi: 10.1093/bja/aeq041. Epub 2010 Mar 5. PMID 20207747
- [Background] Ghanavatian S, James DL, Sadolf JS. The role of short-term, low dose intravenous ketamine infusion in Calciphylaxis. CEN Case Rep. 2021 Aug;10(3):422-425. doi: 10.1007/s13730-020-00557-8. Epub 2021 Feb 19. PMID 33606191
- [Background] Mathews TJ, Churchhouse AM, Housden T, Dunning J. Does adding ketamine to morphine patient-controlled analgesia safely improve post-thoracotomy pain? Interact Cardiovasc Thorac Surg. 2012 Feb;14(2):194-9. doi: 10.1093/icvts/ivr081. Epub 2011 Nov 28. PMID 22159259
- [Background] Javery KB, Ussery TW, Steger HG, Colclough GW. Comparison of morphine and morphine with ketamine for postoperative analgesia. Can J Anaesth. 1996 Mar;43(3):212-5. doi: 10.1007/BF03011736. PMID 8829857